CLINICAL TRIAL: NCT02881346
Title: Prospective, Observational, Non-interventional, Multicenter Study on the Efficacy and Tolerability of Calcipotriol/Betamethasone Aerosol Foam (Enstilar®) in Patients With Plaque Psoriasis Under Daily Practice Conditions
Brief Title: Efficacy and Tolerability of Enstilar® in Daily Practice
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ENSTILAR-1295
Record Dates: First submitted 2016-08-23; First posted 2016-08-29 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis vulgaris; Plaque; Topical; Calcipotriol; Foam; Spray
MeSH Terms: conditions — Plaque, Amyloid | interventions — betamethasone dipropionate, calcipotriol drug combination; calcipotriene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enstilar®: Patients with psoriasis vulgaris plaques on body and/or extremities will apply Enstilar® (calcipotriol /betamethasone dipropionate (50 micrograms/g + 0.5 mg/g) cutaneous foam) once daily for up to 4 weeks, according to the approved labelling of Enstilar® in Germany.
  Interventions: Drug: Enstilar®

INTERVENTIONS:
Drug: Enstilar® — Once daily application of cutaneous foam to plaques on body and/or extremities
  Other Names: calcipotriol/betamethasone dipropionate cutaneous foam

SUMMARY:
This study aims to assess how the Enstilar® aerosol foam performs in daily real-life practice with regards to effectiveness and convenience of application to psoriasis plaques on body and extremities. In addition the profiles of patients prescribed Enstilar® will be described, and preceeding, concomitant and follow-up management will be mapped. The study will be conducted in about 100 dermatology clinics all over Germany,

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Psoriasis vulgaris
* Lesions on trunk and/or extremities of at least mild severity
* Treatment with Enstilar® planned
* Signed informed consent to participate

Exclusion Criteria:

* Enrolled in any interventional clinical trial
* Ongoing or recent treatment with any systemic psoriasis
* Ongoing or recent treatment with UV-therapy
* Ongoing or previous treatment with Enstilar®
* Psoriasis of scalp only
* Other forms of psoriasis, e.g. erythrodermic or pustular psoriasis
* More than 30% of surface area affected by psoriasis
* Any contraindications or known allergies to Enstilar® or its ingredients
* Incapacitated patients under institutionalized care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with psoriasis vulgaris plaques on trunk and/or extremities of at least mild severity for whom topical treatment with Enstilar® is planned
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment | Week 4
  5-point Likert scale
Percentage of total body surface area affected | 4 weeks
  Percentage
Absence of related adverse events (ADR) | 4 weeks
  Proportion of patients with no ADRs

SECONDARY OUTCOMES:
Patient Global Assessment | 4 weeks
  5-point Likert scale
PASI 50 | 4 weeks
  Psoriasis Area and Severity Index
PASI 75 | 4 weeks
  Psoriasis Area and Severity Index
Patient reported itching | 4 weeks
  10-point scale
Patient reported sleep loss | 4 weeks
  10-point scale
Patient reported erythema | 4 weeks
  10-point scale
Patient reported scaling | 4 weeks
  10-point scale
Patient reported dry skin | 4 weeks
  10-point scale
Patient reported overall treatment satisfaction | 4 weeks
  4-point Likert scale
Patient reported satisfaction with effectiveness | 4 weeks
  4-point Likert scale
Patient reported satisfaction with tolerability | 4 weeks
  4-point Likert scale
Patient reported satisfaction with convenience | 4 weeks
  4-point Likert scale
Dermatology Life Quality Index | 4 weeks
  Standard Quality of Life Questionnaire (DLQI)

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Gerdes, Dr.med., Principal Investigator — Clinic for Dermatology, Venereology and Allergy, University Clinic Schleswig-Holstein, Campus Kiel
Locations (1):
- Clinic for Dermatology, Venereology and Allergy, University Clinic Schleswig-Holstein, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langley RG, Feldman SR, Nyirady J, van de Kerkhof P, Papavassilis C. The 5-point Investigator's Global Assessment (IGA) Scale: A modified tool for evaluating plaque psoriasis severity in clinical trials. J Dermatolog Treat. 2015 Feb;26(1):23-31. doi: 10.3109/09546634.2013.865009. Epub 2013 Dec 20. PMID 24354461
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Result] Gerdes S, Krakor M, Anger T, Hutt HJ, Korber A. Prospective, Observational, Non-Interventional, Multicentre Study on the Efficacy and Tolerability of a New Calcipotriol/Betamethasone Aerosol Foam (Enstilar(R)) in Patients with Plaque Psoriasis under Daily Practice Conditions. Dermatology. 2017;233(6):425-434. doi: 10.1159/000486700. Epub 2018 Mar 2. PMID 29502110